CLINICAL TRIAL: NCT06691880
Title: Translating SMARTS 2: the Integration of Video Gaming Technology Into Traditional Rehabilitation
Brief Title: Feasibility of Video Gaming Technology for Arm Recovery Early Post-stroke
Acronym: SMARTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00204731
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Subacute Stroke; Acute Stroke
Keywords: stroke; brain repair; recovery; video gaming; Implementation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video Gaming Technology (VGT) based arm training (Experimental): Patients who meet inclusion criteria will be assessed for level of arm impairment and allocated to either MindPod VGT or Bimanual Arm Trainer VGT based on the severity of impairment. Patients will complete up to 60 minutes of VGT treatment in addition to the standard of care therapy (Physical, occupational, and or speech therapy). Patients will be monitored before, during, and after the sessions for tolerance and response to the treatment. This will include physiological response using measures such as blood pressure, heart rate, and pulse oximeter. Self reported pain and fatigue will be collected using visual analog scales. Safety issues that are predefined as line dislodgement, falls, change in vital signs or pain necessitating interruption of the therapy session will be measured and calculated as the number of adverse events as a proportion of the number of sessions attended
  Interventions: Behavioral: MindPod Dolphin VGT; Behavioral: Bimanual Arm Trainer VGT

INTERVENTIONS:
Behavioral: MindPod Dolphin VGT — The MindPod Dolphin, is an interactive video game that allows users to engage in "non-task-based tasks" to motivate the users to play and relearn motor skills. The MindPod gaming platform uses markerless tracking to sense the patient's affected arm. The paretic limb controls Bandit the dolphin underwater in an effort to eat fish. The patient learns to map his/her movements to Bandit in a 3-Dimensional work space to reach the targets. During gaming, the therapist titrates game difficulty. Bilateral gaming components are used (the participant uses a controller with the participant's less-affected limb to control the timing of Bandit's movement) and in-game difficulty can be adjusted to create an immersive, challenging, and engaging experience. In order to be successful, the patient must coordinate both arms to control the temporal and spatial aspects of the game.
Behavioral: Bimanual Arm Trainer VGT — The bimanual arm trainer (BAT) is a device that involves hardware that interfaces with a computer game. The BAT promotes shoulder external rotation and elbow extension in the paretic arm by coupling movements of the paretic arm with the less affected limb as the participant matches his/her arm movements to those of a virtual avatar. The less-affected side and paretic limb are placed in the BAT apparatus and the less affected limb "drives" the impaired limb through passive, symmetrical movements that simulate rowing down a virtual river. The protocol created by the investigators group, leads the patient through an active-passive training progression similar to paradigms used in neural priming studies. Through these series of movements, the goal is to restore balance between the muscles of the upper back and chest to maximize range of motion in preparation for improved quality of movement.

SUMMARY:
The investigators are investigating ways to incorporate new technologies that can enhance functional outcome after neurological insult into the patient recovery space. In order to accelerate the translation of these technologies to patient care spaces, the investigators need to identify the locations that are feasible for its use. Currently the investigators are using video game technologies that are used to maximize motor recovery of impaired upper extremities after neurological insult in the outpatient (clinic) setting. These technologies interface with robotics and other hardware to create a therapy experience that is fun, engaging, dynamic, challenging, and promotes repetitions that are otherwise difficult to achieve during conventional post-stroke rehabilitation. The investigators think early use of these technologies could enhance recovery of the arm, but It is not known if use of these technologies in the early post-stroke recovery period is safe and feasible.

DETAILED DESCRIPTION:
This study explores a protocolized approach to high-dosed, video-game-based arm training in addition to standard of care rehabilitation in the acute/sub-acute phase of stroke recovery. Patients admitted to the Johns Hopkins Hospital rehabilitation unit or the Brain Rescue Unit with new unilateral upper limb weakness as a result of the patient's sequela will be considered for enrollment. Once consented, participants will be seen 4-5 days per week for up to 60 minutes of additional arm training using gaming technology. Participant response to training will be measured before and after the intervention and function and impairment level will be measured pre and post the training protocol. Participants will be expected to participate in the training protocol for the duration of the hospital stay.

The study involves patients who were already hospitalized at a large teaching institution in Maryland. Participants were screened for eligibility on admission to the hospital. If eligible, the patient was screened in person to determine if he/she was able to follow a 1 step functional command and for willingness to participate. Once agreeable, patients and/or the patient's surrogate decision makers were consented to enroll into the study. Patients were included if a stroke was confirmed by CT or MRI with subsequent unilateral upper extremity weakness (as defined as change in functional use of extremity from baseline or difference in Manual Muscle Testing (MMT) score from unaffected side to affected side). Patients were excluded if unable to sit upright for at least 5 minutes in a chair without arm support, unable to follow 1 step functional commands or had a vision impairment that impeded seeing the television screen. Patients were also excluded if the patient had medical instability as defined by the care provider, orthopedic range of motion precautions including, but not limited to: no active range of motion or weight bearing of the target extremity, heart conditions that limits participation in exercise, active seizures or epilepsy or the inability to communicate pain status.

Once consented, baseline assessments are administered and include the FM-UE and dynamometry. The patients are stratified to a gaming technology based on the baseline FM-UE score. Patients with a FM-UE less than 25 are placed in the Bimanual Arm Training group. During the treatment session, the patients are monitored for tolerance of the session using pre and post vitals including Blood Pressure, Heart Rate, and pulse oximetry. Pre/post pain and fatigue ratings are also maintained using a 10 point-likert scale. Trained clinicians gathered session start and end time. Technological difficulties and other interruptions are documented. Adverse events are gathered and include any swelling or bruising, cut/scratch/irritations, and new numbness or tingling. Intervention clinicians use a detailed stopping criteria to monitor the patient for tolerance and participation in the target time on task. The subjects receive intervention daily outside of the subject's regularly scheduled therapy for the 4-5 days a week (pending clinician availability) for the length of the hospital stay.

On the day of or day prior to discharge, FM-UE and dynamometry is gathered again. Qualitative post-intervention outcome measures are gathered for and included a survey of the patient's experience using a Likert-Scale based questionnaire, a Technology Acceptance Model survey (examines the patient's experience using technology and breaks it down into previously defined domains: Perceived Ease of Use (PEU), Perceived Usefulness (PU), Attitude Toward Using (ATU), Behavioral Intention to Use (BIU), and the Intrinsic Motivation Inventory (IMI).

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to Meyer 7 inpatient rehabilitation unit (CIIRP) or Zayed 12 West (12W) Brain Rescue Unit (BRU)
2. Unilateral upper extremity weakness (as defined as change in functional use of extremity from baseline or difference in MMT score from unaffected side to affected side)

Exclusion Criteria:

1. Unable to sit upright for at least 3 minutes
2. Unable to follow 1 step commands
3. Vision impairment that impedes seeing the television screen
4. Medical instability as defined by the care provider
5. Orthopedic range of motion precautions including, but not limited to: no active range of motion or weight bearing of the target extremity
6. Heart condition that limits participation in exercise
7. Active seizures or epilepsy
8. Inability to communicate pain status

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Adherence to the protocol as assessed by session attendance | Immediately Post Intervention
  Adherence to the protocol will be calculated by determining the number of sessions attended as a proportion of the number of possible sessions.
Feasibility: Efficiency (total time on task) | Immediately Post Intervention
  Efficiency will be calculated by examining the amount of practice (Total time on task) as a proportion of total minutes (Total protocol target duration).
Feasibility: Acceptability of the intervention as assessed by the Technology Acceptance Measure | Post intervention up to 2 weeks
  Technology Acceptance Measure; scale range is 1-7 (Strongly disagree to Strongly agree) and higher scores indicate better acceptability.
Feasibility: Acceptability of the intervention as assessed by the Intrinsic Motivation Inventory | Post Intervention up to 2 weeks
  Acceptability of the intervention will be gathered using the Intrinsic Motivation Inventory. This is a 19-item inventory using a 1-7 scale (not at all true to very true) with 3 sub scales: Interest/Enjoyment, Value/Usefulness, Effort/Importance. Higher scores indicate high acceptability.
Heart rate | Baseline, Immediately Post-Intervention
  Heart rate; mean number of beats per minute.
Blood pressure (mmHg) | Baseline, Immediately Post-Intervention
  Systolic and diastolic blood pressure.
Pain as assessed by Wong-Baker Faces Pain Rating Scale | Baseline, Immediately Post-Intervention
  Pain score; (0-10) 10 indicates high level of pain
Fatigue as assessed by Fatigue Visual Analog Scale | Baseline, Immediately Post-Intervention
  Fatigue score; 0-10 with 10 being greater levels of fatigue
Safety as assessed by the number of adverse events | Baseline, Immediately Post-Intervention
  Safety as assessed by the number of adverse events.

SECONDARY OUTCOMES:
Efficacy: Fugl Meyer Upper Extremity | Baseline, Immediately Post-Intervention
  66-point scale that looks at change in arm and hand function at the impairment level as assessed by the Fugl Meyer Upper Extremity Assessment of motor control (FM-UE). The FM-UE uses a 3-point ordinal scale to evaluate sensorimotor function of the arm and hand of the affected upper extremity during reach and grasp movements in and out of synergistic movement patterns. Total scores of 66 are equal to normal movement or no impairment.
Efficacy: Gross Grasp (Dynamometry) | Baseline, Immediately Post-Intervention
  Change in gross grasp will be captured using dynamometry measured in pounds of force output. Three measures will be taken on the right and left hand and the value will be averaged using a calibrated dynamometer and standardized testing procedure. Greater force output is equal to greater grip strength.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Bahouth, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gladstone DJ, Danells CJ, Black SE. The fugl-meyer assessment of motor recovery after stroke: a critical review of its measurement properties. Neurorehabil Neural Repair. 2002 Sep;16(3):232-40. doi: 10.1177/154596802401105171. PMID 12234086
- [Background] Prabhakaran S, Zarahn E, Riley C, Speizer A, Chong JY, Lazar RM, Marshall RS, Krakauer JW. Inter-individual variability in the capacity for motor recovery after ischemic stroke. Neurorehabil Neural Repair. 2008 Jan-Feb;22(1):64-71. doi: 10.1177/1545968307305302. Epub 2007 Aug 8. PMID 17687024
- [Background] Zeiler SR, Krakauer JW. The interaction between training and plasticity in the poststroke brain. Curr Opin Neurol. 2013 Dec;26(6):609-16. doi: 10.1097/WCO.0000000000000025. PMID 24136129
- [Background] Zeiler SR, Hubbard R, Gibson EM, Zheng T, Ng K, O'Brien R, Krakauer JW. Paradoxical Motor Recovery From a First Stroke After Induction of a Second Stroke: Reopening a Postischemic Sensitive Period. Neurorehabil Neural Repair. 2016 Sep;30(8):794-800. doi: 10.1177/1545968315624783. Epub 2015 Dec 31. PMID 26721868
- [Background] Stanmore E, Stubbs B, Vancampfort D, de Bruin ED, Firth J. The effect of active video games on cognitive functioning in clinical and non-clinical populations: A meta-analysis of randomized controlled trials. Neurosci Biobehav Rev. 2017 Jul;78:34-43. doi: 10.1016/j.neubiorev.2017.04.011. Epub 2017 Apr 23. PMID 28442405
- [Background] Gagnon MP, Orruno E, Asua J, Abdeljelil AB, Emparanza J. Using a modified technology acceptance model to evaluate healthcare professionals' adoption of a new telemonitoring system. Telemed J E Health. 2012 Jan-Feb;18(1):54-9. doi: 10.1089/tmj.2011.0066. Epub 2011 Nov 14. PMID 22082108
- [Background] Aminov A, Rogers JM, Middleton S, Caeyenberghs K, Wilson PH. What do randomized controlled trials say about virtual rehabilitation in stroke? A systematic literature review and meta-analysis of upper-limb and cognitive outcomes. J Neuroeng Rehabil. 2018 Mar 27;15(1):29. doi: 10.1186/s12984-018-0370-2. PMID 29587853
- [Background] Hayward KS, Brauer SG. Dose of arm activity training during acute and subacute rehabilitation post stroke: a systematic review of the literature. Clin Rehabil. 2015 Dec;29(12):1234-43. doi: 10.1177/0269215514565395. Epub 2015 Jan 7. PMID 25568073
- [Background] Morris ZS, Wooding S, Grant J. The answer is 17 years, what is the question: understanding time lags in translational research. J R Soc Med. 2011 Dec;104(12):510-20. doi: 10.1258/jrsm.2011.110180. PMID 22179294